CLINICAL TRIAL: NCT05921487
Title: Time Restricted Eating to Mitigate Obesity in Veterans With Spinal Cord Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B4538-M; 1IK1RX004538-01A1 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury; Obesity
MeSH Terms: conditions — Spinal Cord Injuries; Obesity

STUDY DESIGN:
Intervention Model Description: Intervention: This is a single-arm study in a convenience sample of Veterans with paraplegia and obesity.
  Research Design: Those with mean eating windows of at least 10 hours per day will be eligible to participate in the TRE intervention. Tests for adherence (food log) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Time Restricted Eating (Experimental): This is a single-arm study in a convenience sample of Veterans with paraplegia and obesity. The intervention will test adherence of participants to a TRE window with a self-selected start time. The duration of the eating window will be 10 hours, maintained through study's end (end of week 6).
  Interventions: Behavioral: Time Restricted Eating

INTERVENTIONS:
Behavioral: Time Restricted Eating — Time Restricted Eating Protocol: Subjects will be instructed to limit caloric consumption to a 10-hour TRE window. The window start-time will be self-selected (individualized). During the eating window, subjects will not be restricted on types or quantities of food consumed, and will be advised to continue their usual diets. Subjects will not be required to monitor their caloric intake. During the fasting period, subjects will be encouraged to stay hydrated and drink ample water. Outside the designated eating window, subjects are only permitted to consume medication, water, or zero-calorie herbal drinks such as unsweetened tea or black coffee.
  Other Names: TRE

SUMMARY:
Spinal cord injury (SCI) causes paralysis and muscle atrophy and leads to weight gain and obesity. Obesity directly contributes to functional impairment and cardiometabolic dysfunction. There is a critical need to reduce the growing prevalence of obesity and cardiometabolic disease after SCI. My overall objective in this project is to gather crucial feasibility data on time restricted eating (TRE), a novel form of intermittent fasting. TRE is a straightforward method to induce weight loss without the need for calorie counting. TRE allows individuals to eat all their daily calories in a time restricted window and fast outside that window. A growing body of literature supports the safety and efficacy of TRE. Given the feasibility, high adherence, and substantial benefits of TRE in able-bodied individuals, it is important to test TRE to determine its feasibility in Veterans with SCI. The investigators will first test this intervention in Veterans with paraplegia, who are at greatest risk of muscle-joint upper body injury given the need to support body weight during activity. The investigators will determine adherence to a TRE window for 6-weeks duration in a convenience sample of Veterans with paraplegia and obesity. Based on the expected outcomes of good adherence, this study will lay the groundwork for future work by informing the design of a randomized controlled trial to test the efficacy of TRE to facilitate weight loss and improve function.

ELIGIBILITY:
Inclusion Criteria:

* Veteran, age 18 to 89 years old
* The Syracuse SCI registry includes adults only, so the youngest age of enrollment is 18. The effects of fasting on age-induced sarcopenia remain "uncertain"; therefore, the investigators will cap the age at 89 years old
* A member of the Spinal Cord Injury/Disorder (SCI/D) registry through the Syracuse VA, including both hub and spoke sites
* A qualifying diagnosis of SCI within the SCI/D registry
* Neurologic level of injury from T1 to S5, based on most recent Status Update or ASIA examination, or a diagnosis of a hereditary form of paraplegia (such as familial spastic paraplegia or hereditary spastic paraplegia)
* ASIA Impairment Scale grade A-D
* Chronic SCI (> 1 year from date of SCI or diagnosis of SCI)
* BMI > 22 - the BMI used to diagnose obesity in individuals with SCI
* Mean eating window of at least 10 hours per day

Exclusion Criteria:

* Females who are pregnant (tested via urinary hCG), planning to become pregnant in the next 6 months, or breast-feeding
* A member of the SCI/D registry through the Syracuse VA, with a qualifying diagnosis of MS or ALS
* Diagnosis of heart failure
* Diagnosis of diabetes mellitus, type 1
* Diagnosis of diabetes mellitus, type 2, and on insulin or other antidiabetic agent with high incidence of hypoglycemia

  o Of note, antidiabetic agents with low incidence of hypoglycemia are: metformin, GLP-1 receptor agonists, SGLT2 inhibitors, DPP4 inhibitors, alpha glucosidase inhibitors, thiazolidinediones (as discussed with VA pharmacist)
* Diagnosis of End Stage Renal Disease
* Diagnosis of dementia
* Diagnosis of orthostatic hypotension and prescribed midodrine or fludrocortisone
* History of syncopal episode in the month prior to the study
* History of significant weight loss (> 10% body weight) in the month prior to the study
* History of eating disorders (e.g., anorexia or bulimia) within the last five years, or clearance from a mental health provider
* History of active suicidal ideation in the last six months, or clearance from a mental health provider
* Currently prescribed weight loss medication (e.g., liraglutide)
* Currently prescribed corticosteroids
* Current acute medical issues including cancer, sepsis, advanced liver failure, porphyria, or uncontrolled hyperthyroidism

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the daily eating window | Measured weekly from baseline to week 6
  Measured by questionnaire (assesses the time the participant started and stopped eating each day)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey V Henderson, MD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared upon written request for appropriate scientific reasons.
Supporting Information: SAP
Time Frame: The dataset will be available following publication of the primary manuscript for this project.
Access Criteria: The dataset will be released upon written request for scientific purposes including re-analysis and validation of results.